CLINICAL TRIAL: NCT04993443
Title: A Single and Multiple-dose Escalation First-in-Human Study Evaluating the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of LQ036 Administered Via Inhalation and IV Infusion in Healthy Subjects and Patients With Mild Asthma.
Brief Title: First-In-Human Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of LQ036
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Copmeletion of Part A SAD cohorts, sponsor cancelled Part B-D cohorts
Sponsor: Syneos Health (Other)
Collaborators: Shanghai Novamab Biopharmaceuticals Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LQ036A001
Record Dates: First submitted 2021-05-17; First posted 2021-08-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2021-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Drug :LQ036 (Experimental): Experimental, Single and Multiple Oral escalating dose
  Interventions: Drug: LQ036
- Placebo Comparator: Matching Placebo for LQ036 (Placebo Comparator): Matching Placebo for LQ036: Matching Placebo
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: LQ036 — For Each part of the study, a staggered dosing schedule may be used for the first dose level, in each cohort including 2 sentinel subjects (1 active and 1 placebo) initiating dosing first and the remaining 6 subjects for Part A-C and 8 subjects for Part D initiating dosing no sooner than the next day. Each study part (A, B, C, and D) will be completed sequentially, but with partial overlapping. Part B and C may only be initiated after review of the safety, tolerability, and PK data following dosing of the SAD Cohort 3 or 4.
  Part D may be initiated when safety tolerability and PK data are known and deemed acceptable by the SRC for multiple doses in Part B, at least at the same concentration to be administered in Part D.
  Arms: Active Comparator: Drug :LQ036
Other: Matching Placebo — Matching Placebo for LQ036: Matching Placebo
  Other Names: Matching Placebo for LQ036
  Arms: Placebo Comparator: Matching Placebo for LQ036

SUMMARY:
This is Phase I first-in-human trial evaluating the safety, tolerability, immunogenicity, and pharmacogenomics of LQ036 via inhalation and IV infusion.

The study will be divided into 4 parts: Single Ascending Dose, Multiple Ascending Dose, and Intra Venous with a target of 88 healthy volunteers and 30 patients with mild Asthma.

DETAILED DESCRIPTION:
This study will be a Multicenter, phase Ia/Ib, randomized, double-blind, placebo controlled, Single Ascending Dose(SAD)/ Multiple Ascending Dose (MAD) study of dose escalation cohorts evaluating the safety, tolerability, immunogenicity, and PK of LQ036 after administration via inhalation and intravenous (IV) infusion in healthy subjects and patients with mild Asthma.

The study will be divided into 4 parts:

The four parts will be completed sequentially or with partial overlapping.

Part A - SAD Cohorts (A1 to A5):

A staggered dosing schedule will be followed, for each cohort: 2 sentinel subjects (1 active and 1 placebo) will be dosed and the remaining 6 subjects will be dosed no sooner than the next day.

Cohorts will be dosed sequentially in an ascending fashion. There will be at least 14 days between dosing of each dose level. Following completion of each dose level, a safety review committee (SRC) composed by at least the Investigator, a Sponsor representative, and an Independent Medical monitor will review the safety and tolerability data, as well as available PK and immunogenicity data up to Day 15, for at least 6 subjects in the respective cohort, as well as available PK and immunogenicity data. Decisions from the SRC may include whether to escalate to the next dose level, continue with a more conservative approach (slowing the increase in dose or repeating a dose level), suspending dose escalation until further review of study data, stopping dose escalation, or terminating the study.

Part B - MAD Cohorts (B1 to B4):

Part B can be initiated only following review of the safety, tolerability, and PK data following dosing of the SAD Cohort 3 or 4, if deemed acceptable by the SRC.

A staggered dosing schedule may be used for the first dose level, including 2 sentinel subjects (1 active and 1 placebo) initiating dosing first and the remaining 6 subjects initiating dosing no sooner than the next day.

Cohorts will be dosed sequentially in an ascending fashion. There will be at least 14 days between dosing of each dose level. Following completion of each dose level, a SRC composed of at least the Investigator, a Sponsor representative, and an Independent Medical monitor will review the safety and tolerability data up to Day 15, for at least 6 subjects in the respective cohort, as well as available PK and immunogenicity data.

Decisions from the SRC may include whether to escalate to the next dose level, continue with a more conservative approach (slowing the increase in dose, repeating a dose level, or exploring an alternative dosing regimen), suspending dose escalation until further review of study data, stopping dose escalation, or terminating the study.

Part C - IV Cohorts (C1 and C2):

Part C can be initiated only following review of the safety, tolerability, and PK data following dosing of the SAD Cohort 3 or 4, if deemed acceptable by the SRC.

A staggered dosing schedule will be followed for each cohort: 2 sentinel subjects (1 active and 1 placebo) will be dosed first and the remaining 6 subjects will be dosed no sooner than the next day.

Cohorts will be dosed sequentially in an ascending fashion. There will be at least 14 days between dosing of each dose level. Following completion of each dose level, The SRC composed by at least the Investigator, a Sponsor representative, and an Independent Medical monitor will review the safety and tolerability data up to Day 15, for at least 6 subjects in the respective cohort, as well as available PK and immunogenicity data. Decisions from the SRC may include whether to escalate to the next dose level, continue with a more conservative approach (slowing the increase in dose or repeating a dose level), suspending dose escalation until further review of study data, stopping dose escalation, or terminating the study.

Some alterations from the currently outlined dose and/or dosing regimen may be performed, but the dose to be administered in a given cohort will not exceed the one currently outlined in the protocol.

Part D (Multiple Dose Patients) - Cohorts D1 to D3:

Part D may be initiated following submission and review of an interim analysis report from Parts A through C of the study by both the SRC and Human Research Ethics Committee (HREC). Part D may commence only after approval to commence from both committees is granted.

A staggered dosing schedule may be used for each cohort. Two (2) sentinel subjects (1 active and 1 placebo) will initiate dosing first (a minimum of 1 hour apart from end of dosing for first sentinel patient to start of dosing for second sentinel patient) and the remaining 8 subjects will initiate dosing no sooner than the next day (each dosed at least 15 minutes apart from end of dosing for previous patient to start of dosing for following patient). Cohorts will be dosed either sequentially or with partial overlapping and the SRC will meet to discuss relevant data collected after completion of at least the first cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as defined by:

  1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
  2. the absence of a clinically significant history of neurological, endocrine, cardiovascular, respiratory (except resolved childhood asthma), hematological, immunological, psychiatric (except including depression that has not required treatment for at least 6 months), gastrointestinal, renal, hepatic, and metabolic disease.
* Male or female, non-smokers or casual smokers (defined as smoking the equivalent of less than an average of 5 cigarettes per week over a 3 month period, and willing to abstain from smoking during involvement in the study and for 1 month prior to screening), ≥18 and ≤55 years of age, with BMI >18.0 and <32.0 kg/m2.
* Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:

  1. Simultaneous use of intrauterine device placed at least 4 weeks prior to study drug administration, and condom for the male partner;
  2. Simultaneous use of hormonal contraceptives started at least 4 weeks prior to study drug administration and condom for the male partner.
  3. Sterile male partner (vasectomized since at least 6 months).
* Male subjects who are sexually active with a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must be willing to use one of the following acceptable contraceptive methods from the first study drug administration until at least 90 days after the last study drug administration:

  1. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives used since at least 4 weeks, or intra-uterine contraceptive device placed since at least 4 weeks;
  2. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
* Subjects with normal lung function defined as greater than or equal to 80% predicted forced expiratory volume in one second (FEV1).
* Males and females who are in same-sex relationships can be included. There are no mandatory contraceptive requirements for males or females in same-sex relationships.
* Male and female heterosexual subjects who practice abstinence from sexual intercourse as a usual and preferred lifestyle.
* Part D only: Volunteers with mild asthma defined as:

  1. Asthma diagnosed with appropriate medical documentation;
  2. FEV1 ≥70% predicted FEV1 and FEV1/FVC ratio ≥0.7 at screening;
  3. FeNO ≥35 ppb at screening;
  4. Well-controlled, or partly-controlled, by as-needed use of short-acting β2 agonists for at least 3 months prior to dosing;
  5. Reversibility test at screening consistent with diagnosis of asthma (≥12% and 200 mL increase in FEV1 over the baseline value).
* Capable of consent

Exclusion Criteria:

* Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C found at screening or at check-in (Day -1, not applicable to serology assessments).
* Any clinically significant illness, infection, medical/surgical procedure, or trauma within 4 weeks of check-in, or planned inpatient surgery or hospitalization during the study period.
* Any history of malignancy or neoplastic disease (not including excised, non-recurrent, non-melanoma skin cancers).
* Positive urine drug screen, urine cotinine test, or alcohol breath test at screening or at check-in (Day -1).
* History of allergic reactions to LQ036, to any biologic therapy, or other related drugs, or to any excipient in the formulation.
* Positive pregnancy test at screening or at check-in (Day -1)
* Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure less than 90 or greater than 140 mmHg, diastolic blood pressure less than 40 or greater than 90 mmHg, or heart rate less than 40 or greater than 100 bpm) at screening.
* History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit. Regular use of alcohol is defined as greater than 14 units of alcohol per week, where 1 unit is defined as 100 mL of wine at 13.5% a/v, 375 mL of beer at 3.5% a/v, or 30 mL of spirit at 40% a/v.
* History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as tetrahydrocannabinol) within 1 month prior to the screening visit or hard drugs (amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine, and phencyclidine) within 3 months prior to screening.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
* Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

  1. Prescription medications (except for hormonal contraceptives in all study parts and short-acting β2 agonists for patients in Part D) within 14 days prior to the first dosing;
  2. Over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing, with the exception of the occasional use of paracetamol/acetaminophen (up to 2 g daily), ibuprofen (up to 800 mg daily), and oral contraceptives;
  3. Depot injection or implant (except for hormonal contraceptives) of any drug within 3 months prior to the first dosing;
  4. Long-acting ß2 agonists for 4 weeks prior to screening;
  5. Anti-immunoglobulin E,anti-Interleukin-5, or anti-Interleukin-4 Receptor therapy for 6 months prior to screening;
  6. Inhaled corticosteroids (greater than 500 μg/day of beclometasone dipropionate or equivalent) within 16 weeks prior to screening,
  7. Oral or injectable steroids for the treatment of asthma or respiratory tract infection within 5 years prior to screening;
  8. Intranasal steroids within 4 weeks prior to screening;
  9. Topical steroids within 4 weeks prior to screening;
  10. Leukotriene antagonists within 2 weeks prior to screening;
  11. Anticholinergics or cromoglycate within 1 week prior to screening.
  12. Inhaled short-acting β2 agonists (such as salbutamol) within 6 months prior to screening (not applicable to patients in Part D).
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
* Breast-feeding subject.
* History of latent or active tuberculosis, or exposure to endemic areas within 8 weeks prior to QuantiFERON®-TB testing performed at screening.
* Positive QuantiFERON®-TB test indicating possible tuberculosis infection.
* Immunization with a live attenuated vaccine within 1 month prior to dosing or planned vaccination during the course of the study.
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening.
* History of clinically significant opportunistic infection (e.g., invasive candidiasis or one pneumocystis pneumonia).
* History of parasitic diseases (e.g., toxoplasmosis, cysticercosis, toxocariasis).
* History of frequent, recurrent herpes simplex.
* Presence of fever (body temperature greater than 37.6 °C) e.g., a fever associated with a symptomatic viral or bacterial infection, within 2 weeks prior to the first dosing.
* Life threatening asthmatic episode at any time in the past.
* C-reactive protein level above 5 mg/L.
* Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 weeks.
  Assessment of outcome of Adverse events
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 1 Month
  Abnormal blood pressure
  Part A and C: At check-in (Day -1), pre-dose (Day 1), and 1, 2, 4, 6, 8, 12, and 24 (Day 2) hours post-dose, at discharge (Day 3), and on Days 8±1, 15±1, and 22±1.
  Part B and D: At check-in (Day -1), on Day 1: pre-dose, and 1, 2, 4, 6, 8, and 12 hours-post first dose, pre-dose and 2 and 6 hours post-dose on Days 2 to 10, and on Days 11, 12, 13, 15±1, 22±1, and 29±1.
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 1 Month
  Abnormal pulse rate
  Part A and C: At check-in (Day -1), pre-dose (Day 1), and 1, 2, 4, 6, 8, 12, and 24 (Day 2) hours post-dose, at discharge (Day 3), and on Days 8±1, 15±1, and 22±1.
  Part B and D: At check-in (Day -1), on Day 1: pre-dose, and 1, 2, 4, 6, 8, and 12 hours-post first dose, pre-dose and 2 and 6 hours post-dose on Days 2 to 10, and on Days 11, 12, 13, 15±1, 22±1, and 29±1.
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 1 Month
  Abnormal respiratory rate
  Part A and C: At check-in (Day -1), pre-dose (Day 1), and 1, 2, 4, 6, 8, 12, and 24 (Day 2) hours post-dose, at discharge (Day 3), and on Days 8±1, 15±1, and 22±1.
  Part B and D: At check-in (Day -1), on Day 1: pre-dose, and 1, 2, 4, 6, 8, and 12 hours-post first dose, pre-dose and 2 and 6 hours post-dose on Days 2 to 10, and on Days 11, 12, 13, 15±1, 22±1, and 29±1.
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 1 Month
  Abnormal Tympanic Temperature
  Part A and C: At check-in (Day -1), pre-dose (Day 1), and 1, 2, 4, 6, 8, 12, and 24 (Day 2) hours post-dose, at discharge (Day 3), and on Days 8±1, 15±1, and 22±1.
  Part B and D: At check-in (Day -1), on Day 1: pre-dose, and 1, 2, 4, 6, 8, and 12 hours-post first dose, pre-dose and 2 and 6 hours post-dose on Days 2 to 10, and on Days 11, 12, 13, 15±1, 22±1, and 29±1.
To assess changes in cardiovascular system function (change in QTC parameters) as a criterion of safety and tolerability variables. | Up to 1 Month
  Change in electrocardiograms (ECGs).
  Part A and C: At check-in (Day -1), pre-dose (Day 1), and 1, 2, 8, and 24 (Day 2) hours post-dose, at discharge (Day 3), and on Days 8±1, 15±1, and 22±1.
  Part B and D: At check-in (Day -1), and pre-dose and 1, 2, and 8 hours post-dose on Days 1 to 12, and at discharge (Day 13), and on Days 15±1, 22±1, and 29±1.
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (hemoglobin)
  Part B and D: At screening, at check-in (Day -1), on Days 2 and 7, at discharge (Day 13), and at study exit (Day 36±1).
  Part A and C: At screening, at check-in (Day -1), on Day 2, at discharge (Day 3), on Day 8±1, and at study exit (Day 29±1).
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (hematocrit)
  Part B and D: At screening, at check-in (Day -1), on Days 2 and 7, at discharge (Day 13), and at study exit (Day 36±1).
  Part A and C: At screening, at check-in (Day -1), on Day 2, at discharge (Day 3), on Day 8±1, and at study exit (Day 29±1).
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (mean corpuscular volume)
  Part B and D: At screening, at check-in (Day -1), on Days 2 and 7, at discharge (Day 13), and at study exit (Day 36±1).
  Part A and C: At screening, at check-in (Day -1), on Day 2, at discharge (Day 3), on Day 8±1, and at study exit (Day 29±1).
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (leukocyte counts)
  Part B and D: At screening, at check-in (Day -1), on Days 2 and 7, at discharge (Day 13), and at study exit (Day 36±1).
  Part A and C: At screening, at check-in (Day -1), on Day 2, at discharge (Day 3), on Day 8±1, and at study exit (Day 29±1).
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (platelet count)
  Part B and D: At screening, at check-in (Day -1), on Days 2 and 7, at discharge (Day 13), and at study exit (Day 36±1).
  Part A and C: At screening, at check-in (Day -1), on Day 2, at discharge (Day 3), on Day 8±1, and at study exit (Day 29±1).
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (Urea)
  Part B and D: At check-in (Day -1), on Days 2 and 7, at discharge (Day 13), and at study exit (Day 36±1).
  Part A and C: At screening, at check-in (Day -1), on Day 2, at discharge (Day 3), on Day 8±1, and at study exit (Day 29±1).
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (creatinine)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (alkaline phosphatase)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (glucose)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (alanine aminotransferase (ALT))
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (aspartate amino transferase (AST))
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (total bilirubin)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (sodium)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (potassium)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (chloride)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (calcium)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (total proteins)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (Phosphorus)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (albumin)
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (Coagulation test (aPTT (Activated partial thromboplastin time) and INR (International Normalized Ratio))
  Part B and D: At screening and at study exit (Day 36±1)
  Part A and C: At screening and at study exit (Day 29±1).
To evaluate the safety of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Assessment of abnormal clinical laboratory tests (Urine macroscopic examination, pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, nitrite, urobilinogen, and leukocytes)
  Part B and D: At screening, at check-in (Day -1), on Days 2 and 7, at discharge (Day 13), and at study exit (Day 36±1).
  Part A and C: At screening, at check-in (Day -1), on Day 2, at discharge (Day 3), and at study exit (Day 29±1).
To evaluate the tolerability of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 weeks
  Local tolerability (oropharyngeal) assessment (Part A) and (injection site) assessment (Part C): The area where the study drug was administered will be monitored by study personnel throughout the study for any signs of local reactions such as swelling or redness.
  Time frame: pre-dose, Day 1, 2, 4, 8, and 24 hours post-dose, and at Day 3.
  Local tolerability (oropharyngeal) assessment (Part B and D): The area where the study drug was administered will be monitored by study personnel throughout the study for any signs of local reactions such as swelling or redness.
  Time frame: pre-dose (as well as 1, 2, and 4 hours post-dose on Days 1, 3, 5, 8, and 10, 11, 13, and at day 36.
To evaluate the immunogenicity of single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 5 Weeks
  Immunogenicity data that will be evaluated include Anti-Drug Antibody test sampling (ADA).
  Parts A and C: A total of 5 blood samples will be taken for ADA assessment: at pre-dose (Day 1), and on Days 8±1, 15±1, and 22±1, and at study exit (Day 29±1)
  Part B and D: A total of 6 blood samples will be taken for ADA assessment: at pre-dose (Day 1), and on Days 8±1, 15±1, 22±1, 29±1, and at study exit (Day 36±1)
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects. | Up to 2 Weeks
  AUC0-t: Area under the concentration-time curve from time zero until the last observed concentration
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects. | Up to 2 Weeks
  AUC0-inf: Area under the concentration-time curve from time zero to infinity (extrapolated)
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects. | Up to 2 Weeks
  Residual area: Percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity, calculated as [1 - (AUC0-t/AUC0-inf)] x 100
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  AUC0-24: Area under the concentration-time curve from time zero to 24 hours post-dose.
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  AUC0-τ: Area under the concentration-time curve for one dosing interval (τ) at steady-state. In this study τ = 24 hours (AUC0-24)
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  AUC0-72: Area under the concentration-time curve from time zero to 72 hours post-dose.
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  Cmax: Maximal observed concentration
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  Cmax ss: maximum observed concentration at steady-state
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  Cmin ss: minimum observed concentration at steady-state
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  Tmax ss: time of observed Cmax at steady-state
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  Tmax: Time of Cmax
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects | Up to 2 Weeks
  T½ el: Terminal elimination half-life
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects (Kel) | Up to 2 Weeks
  Kel: Terminal elimination rate constant
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma (Racc) | Up to 2 Weeks
  Racc: drug accumulation ratio
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. (PTF%) | Up to 2 Weeks
  PTF%: peak trough fluctuation
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects. | Up to 2 Weeks
  Cl/F: Apparent body clearance, calculated as Dose / AUC0-inf
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects | Up to 2 Weeks
  Vd/F: apparent volume of distribution, calculated as Dose / Kel * AUC0-inf
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  Clss/F: apparent body clearance at steady-state, calculated as dose / AUC0-inf
To evaluate the pharmacokinetics (PK) of LQ036 after single and multiple doses of LQ036 administered via inhalation and IV routes in healthy subjects and patients with mild Asthma. | Up to 2 Weeks
  Vdss/F: apparent volume of distribution at steady-state, calculated as dose / (Kel * AUC0-inf)
To evaluate the change in fraction exhaled nitric oxide (FeNO) after multiple doses of LQ036 administered via inhalation in patients with mild asthma. | Up to 6 weeks
  At screening, on dosing days (Days 1 to 10, within 60 minutes prior to dosing), on Days 11, 12, and at discharge (Day 13), as well as on Days 15±1, 22±1, 29±1, and at study exit (Day 36±1).

SECONDARY OUTCOMES:
To compare the PK of LQ036 after administration via inhalation and IV routes | Up to 2 weeks
  Serum levels of LQ036 will be quantified for PK analysis by a validated enzyme linked immunosorbent assay (ELISA) method.
To compare the safety and tolerability of LQ036 after administration via inhalation and IV routes (AUC0-24 versus AUC0-τ) | Up to 2 weeks
  Comparisons between Day 1 and Day 10 PK parameters: AUC0-24 versus AUC0-τ will be done by Analysis of variance (ANOVA)
To compare the safety and tolerability of LQ036 after administration via inhalation and IV routes (Cmax versus Cmax ss) | Up to 2 weeks
  Comparisons between Day 1 and Day 10 PK parameters: Cmax versus Cmax ss will be done by Analysis of variance (ANOVA)
To compare the safety and tolerability of LQ036 after administration via inhalation and IV routes (Tmax versus Tmax ss) | Up to 2 weeks
  Comparisons between Day 1 and Day 10 PK parameters: Tmax versus Tmax ss will be done by Analysis of variance (ANOVA)
To compare the PK of LQ036 after administration via inhalation in healthy subjects versus patients with mild asthma. | Up to 2 weeks
  Serum levels of LQ036 will be quantified for PK analysis by a validated enzyme linked immunosorbent assay (ELISA) method
To compare the safety and tolerability of LQ036 via inhalation in healthy subjects versus patients with mild asthma. (AUC0-24 versus AUC0-τ) | Up to 2 weeks
  Comparisons between Day 1 and Day 10 PK parameters: AUC0-24 versusAUC0-τ will be done by Analysis of variance (ANOVA)
To compare the safety and tolerability of LQ036 via inhalation in healthy subjects versus patients with mild asthma. (Cmax versus Cmax ss) | Up to 2 weeks
  Comparisons between Day 1 and Day 10 PK parameters: Cmax versus Cmaxss will be done by Analysis of variance (ANOVA)
To compare the safety and tolerability of LQ036 via inhalation in healthy subjects versus patients with mild asthma. (Tmax versus Tmax ss) | Up to 2 weeks
  Comparisons between Day 1 and Day 10 PK parameters: Tmax versus Tmaxss will be done by Analysis of variance (ANOVA)

CONTACTS AND LOCATIONS:
Overall Officials: Huaiyu Gu, Study Chair — Shanghai Novamab Biopharm Co., Ltd.
Locations (2):
- Australia (2):
  - Q-Pharm Pty Ltd (Nucleus Network Brisbane), Brisbane, Queensland
  - Nucleus Network Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No